CLINICAL TRIAL: NCT04043637
Title: Complete Puborectalis, Puboperinealis Muscle and Urethral Rhabdomyosphincter Preservation in Laparoscopic Radical Prostatectomy: Anatomic Landmarks to Achieving Early Urinary Continence
Brief Title: Early Urinary Continence After Radical Prostatectomy: Surgical Procedure and Anatomic Landmarks
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Other Study IDs: 19/24
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Prostatic Cancer; Surgical Procedure, Unspecified; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study describes how to perform a correct prostatic apex and membranous urethra in order to preserve all anatomical elements that are necessary to achieve a very fast urinary continence after open/laparoscopic/robotic radical prostatectomy, avoiding positive surgical margins at this level.

DETAILED DESCRIPTION:
This study describes a simple technical variation, aimed at the sparing of the muscle systems and neurovascular bundles in order to achieve high rates of urinary continence in the early postoperative period ( the first two months after surgery) in prostate cancer patients undergoing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years
* A Body Mass Index lower than 35 Hg/m2
* Patients with organ-confined prostate cancer
* Signed informed consent

Exclusion Criteria:

* Contraindications for Laparoscopy

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A series of 120 consecutive prostate cancer patients who underwent Laparoscopic Radical Prostatectomy from 2012 to 2018, always performed by the same surgeon
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
change in the proportion of patients with of urinary incontinence | The follow-up was at 2 weeks, 4 weeks and 8 weeks after removal of the urethral catheter (one week after surgery), and, thereafter, once a month over the first year after surgery
  Assessment of the proportion of patients with urinary incontinence after laparoscopic radical prostatectomy

SECONDARY OUTCOMES:
change in the proportion of patients with recovery of the erectile function | every month during the first year after surgery
  assessment of the recovery of the erectile function after surgery
number of patients with overall positive surgical margins | immediate postoperative period
  postoperative assessment of positive surgical margins
biochemical recurrence rate | until the completion of the study, with a mean follow-up of 72 months